CLINICAL TRIAL: NCT01266681
Title: Amiodarone Compared to Dronedarone , Post Cardioversion Maintenance of Sinus
Brief Title: Amiodarone Compared to Dronedarone , Post Cardioversion Maintenance of Sinus Rhythm
Acronym: ACDC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Dr Steven Furniss, East Sussex Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACDC MainS
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiodarone (Active Comparator): this group will be given Amiodarone to maintain sinus rhythm powst cardioversion.
  Interventions: Drug: amiodarone
- Dronedarone (Active Comparator): this group will be given dronedarone to maintain sinus rhythm post DC cardioversion
  Interventions: Drug: Dronedarone

INTERVENTIONS:
Drug: amiodarone — Visit One:. Once consent is given patarticipants will be randomised into either group and instructed and prescribed the drug as appropriate.
  Visit Two: Patients will attend for routine cardioversion. This is performed by an experienced CCU nurse as per normal protocol. Patients will also undergo an ECG, and fill in symptom and quality of life (QoL) questionnaires.
  Visit Three: Patients will attend a routine outpatient appointment 6 weeks post cardioversion. They will undergo ECG and fill in symptom and QoL questionnaires
  Visit Four: Participants will attend at 12 weeks for ECG, symptom and QoL questionnaires
  Visit Five: Participants will attend at 24 weeks for ECG, symptom and QoL questionnaires
  Visit Six: Participants will attend at 36 weeks for ECG, symptom and QoL questionnaires
  Visit Seven: Participants will attend at 52 weeks for ECG, symptom and QoL questionnaires. Participants will then be followed up as per protocol by their consultant cardiologist.
  Arms: Amiodarone
Drug: Dronedarone — Visit One: patarticipants will be randomised into either group and instructed and prescribed the drug as appropriate.
  Visit Two: Patients will attend for routine cardioversion. This is performed by an experienced CCU nurse as per normal protocol. Patients will also undergo an ECG, and fill in symptom and quality of life (QoL) questionnaires.
  Visit Three: Patients will attend a routine outpatient appointment 6 weeks post cardioversion. They will undergo ECG and fill in symptom and QoL questionnaires
  Visit Four: Participants will attend at 12 weeks for ECG, symptom and QoL questionnaires
  Visit Five: Participants will attend at 24 weeks for ECG, symptom and QoL questionnaires
  Visit Six: Participants will attend at 36 weeks for ECG, symptom and QoL questionnaires
  Visit Seven: Participants will attend at 52 weeks for ECG, symptom and QoL questionnaires. Participants will then be followed up as per protocol by their consultant cardiologist.
  Arms: Dronedarone

SUMMARY:
Persistent Atrial Fibrillation (AF) is a common and distressing cardiac arrhythmia and accounts for 1% of the healthcare budget in the UK and it's prevalence is rising. Symptoms of atrial fibrillation include palpitations, chest pain , shortness of breath and fatigue, with quality of life measures reduced for patients with persistent AF, increased stroke risk and increased all cause mortality rates. DC Cardioversion is used to restore normal sinus rhythm in patients with persistent AF. It has a high success rate but reoccurence of AF is common. The use of anti arrhythmic drugs (AADs) can augment the number of patients remaining in sinus rhythm at one year, with amiodarone currently the most superior. Unfortunately it can have serious side affects. Dronedarone is a related drug designed specifically to minimise the most serious side affects and is no approved and used prominently in the management of non permanent AF. However it has not yet been studied in a post DC Cardioversion population.

Patients in persistent AF who are referred for elective DC Cardioversionwill be randomised to receive either Amiodarone or Dronedarone to compare the ability to help maintain sinu rhythm post cardioverion in one NHS hospital. Patients will be followed up for a year post cardioversion to see if they stay in sinus rhythm.

Ho: there will be no difference in maintenance of sinus rhythm with the use of amiodarone or dronedarone

ELIGIBILITY:
Inclusion Criteria:

* • Patients with persAF requiring dc cardioversion.

  * Patients must be over 18 years old.
  * Patients give informed consent form prior to participating in this study.
  * Patients must be on warfarin for at least 4 weeks or a transoesphageal ECHO must be performed at the time of dc cardioversion.

Exclusion Criteria:

* • Patient is suffering with unstable angina in last 1 week.

  * Patient has had a myocardial infarction within last 2 months.
  * Patient is expecting or has had major cardiac surgery within last 2 months.
  * Patient is participating in a conflicting study.
  * Patient is mentally incapacitated and cannot consent or comply with follow-up.
  * Patient has NYHA class III/ IV heart failure.
  * Pregnancy.
  * Patient suffers with other cardiac rhythm disorders.
  * Recent coronary artery intervention or other factors suggesting clinical instability (ECG, clinical or laboratory findings).
  * GFR<30mls/min.
  * Patients has a contraindication to amiodarone or dronedarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
maintenance of sinus rhythm at one year post DC Cardioversion | 1 year

SECONDARY OUTCOMES:
tolerability of amiodarone compared to dronedarone | 1 year
measures of quality of life and symptoms in amiodarone compared to dronedarone | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Eastbourne General Hospital, Eastbourne, East Sussex, United Kingdom